CLINICAL TRIAL: NCT04026542
Title: Factors Associated With Normal Exercise Capacity in Patients With Single Ventricle: the Multicenter Cross-sectional Study
Brief Title: Factors Associated With Normal Exercise Capacity in Patients With Single Ventricle
Acronym: SV
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Collaborators: M3C (complex congenital heart disease) French Network (Unknown)
Responsible Party: Sponsor
Other Study IDs: RECHMPL19_0330
Record Dates: First submitted 2019-07-17; First posted 2019-07-19 (Actual); Last update posted 2021-05-19 (Actual); Status verified 2020-03

CONDITIONS: Univentricular Heart
Keywords: VO2max; Fontan; Congenital heart disease; Single ventricle
MeSH Terms: conditions — Univentricular Heart; Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The congenital heart disease (CHD) is the firts cause of congenital birth defects. Medical and surgical advances completely changed the epidemiology of CHD. Among these CHD, the univentricular heart, or single ventricle (SV), is a disease whose medical-surgical progress has completely changed the epidemiology.

The SV at birth receives systemic and pulmonary venous returns in the single functional cavity and provides systemic and pulmonary flow. The SV undergoes a severe volumetric overload and considerably increases its work, which is not viable for the long time.

In 1968, Professor Francis Fontan created the palliative surgery of the univentricular heart. It consists in establishing a derivation of the systemic venous blood from the two vena cava veins directly to the pulmonary arteries, without a sub-pulmonary ventricle. So, the VU no longer undergoes volumetric overload, and eliminates cyanosis.

In this "Fontan circulation", there is no pump to push the blood in the pulmonary arteries, only the remaining systemic post-capillary energy (reflection of the central venous pressure) allows to drive the blood through the lungs with a risk of stasis upstream (right overload) and a limited pre-charge downstream, which can lead to severe consequences: limited exercise capacity, systolic and diastolic dysfunction of the SV, arrhythmia, cyanosis, cirrhosis and hepatic carcinoma, exudative enteropathy , plastic bronchitis, venous thromboses, deaths.

There is a great heterogeneity within this family of SV with extremely varied evolutionary profiles. The cardiorespiratory exercise test, which has become a "gold standard", makes it possible to assess the severity of CHD. In our study on the aerobic fitness of children with CHD, the investigators found that 44% of children with SV had normal aerobic fitness (> 80% of the theoretical VO2max)1. Some good prognostic criteria are already described: left SV, good VU function, total cavopulmonary shunt in young age, etc. But the investigators know that these elements are not enough to explain why some SV, which the investigators will call the "great-SV", have a better aerobic fitness.

The main objective of our study is to describe the population of "great SV" (VO2max ≥ 80%) within the general population of SV. The investigators thus wish to determine the prognostic criteria favorable to a good aerobic fitness in univenticular heart disease.

DETAILED DESCRIPTION:
This study is cross-sectionnal, multicentric national (M3C network), descriptive, observational.

Children ≥ 6 years old and adults with a single ventricle according to the international classification ACC-CHD and who had a cardiopulmonary exercise test in the year during usual follow-up will be included. Patients refuse the use of medical data will be excluded.

The main objective of our study is to describe the rate of "great SV" (VO2max ≥ 80%) within the general population of SV. The secondary objectives are to compare the two groups: group "great SV" with VO2max ≥ 80% versus group SV with VO2max < 80%.

The following criteria will be collected

Anatomical : left SV, right SV, undetermined SV, total cavopulmoary shunt, partial cavopulmonary shunt

Clinic: NYHA status, saturation, medical treatment, number of surgery procedure, number of catheterization procedure, presence of pacemaker or implantable defibrillator, presence of arrythmia.

Morbidity: number oh hospitalization during the year, presence of arrhythmia, cirrhosis and hepatic carcinoma, exudative enteropathy , plastic bronchitis, venous thromboses, stroke.

Echocardiography: ejection fraction of SV, 2D Strain of SV, atrioventricular valve regurgitation, aortic stenosis, aspect of the flow in the cavopulmonary shunt.

Cardiac MRI: ejection fraction of SV

Cardiac catheterization: mean pulmonary arterial pressure, pulmonary arterial wedge pressure, presence of fistulae.

Cardiopulmonary exercise test : VO2max, anaerobic threesold, VE/VCO2 slope, oxygen uptake efficiciency slope, maximal heart rate, oxygene pulse and saturation at exercise.

Pulmonary functional test : forced expiratory volume in 1 seconde (FEV1), the forced vital capacity (FVC), the FEV1/FVC ratio (FEV1/FVC%), DLCO and residual volume.

ELIGIBILITY:
Inclusion criteria:

- Children ≥ 6 years old and adults with a single ventricle according to the international classification ACC-CHD and who had a cardiopulmonary exercise test in the year during usual follow-up.

Exclusion criteria:

- Patients refuse the use of medical data will be excluded.

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with a single ventricle according to the international classification ACC-CHD who had a cardiopulmonary exercise test in the year during usual follow-up.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
rate of "great SV" (VO2max ≥ 80%) within the general population of SV | 1 day
  * measurement of the VO2max at the annual cardiopulmonary exercise test.
  * rate of patient who have a VO2max ≥ 80% in this population of SV recruited.

SECONDARY OUTCOMES:
Comparison of the 2 groups: "great SV" versus others SV. | 1 day
  Multivariate analysis with the following data to define parameters associated with "great SV": Anatomical, Clinic, Morbidity, Echocardiography, Cardiac MRI, Cardiac catheterization, Cardiopulmonary exercise test, Pulmonary functional test

CONTACTS AND LOCATIONS:
Overall Officials: Arthur GAVOTTO, MD, Principal Investigator — University Hospital, Montpellier; Pascal AMEDRO, MD, PhD, Study Director — University Hospital, Montpellier
Locations (1):
- Uh Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC